CLINICAL TRIAL: NCT04612725
Title: A Phase 2b Multinational, Randomised, Double-blind, Parallel- Group, 24-week Placebo-controlled Study With 28-week Extension to Investigate the Use of Benralizumab in Patients With Chronic Spontaneous Urticaria Who Are Symptomatic Despite the Use of Antihistamines (ARROYO)
Brief Title: A Study to Investigate the Use of Benralizumab in Patients With Chronic Spontaneous Urticaria Who Are Symptomatic Despite the Use of Antihistamines (ARROYO)
Acronym: ARROYO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not meet primary endpoint
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3259C00001; 2020-000169-17 (EudraCT Number)
Record Dates: First submitted 2020-09-18; First posted 2020-11-03 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: chronic spontaneous urticaria,; skin lesion,; pruritus and wheals
MeSH Terms: conditions — Chronic Urticaria; Pruritus; Urticaria | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Benralizumab Arm 1 (Experimental): Benralizumab Dose A regimen A until Week 12, Dose B regimen A until Week 24, and Dose B regimen B during the extension period until Week 52 (n=30)
  Interventions: Biological: Benralizumab
- Benralizumab Arm 2 (Experimental): Benralizumab Dose A regimen A until Week 12, Dose B regimen A until Week 24,and Dose B regimen A during the extension period until Week 52 (n=30)
  Interventions: Biological: Benralizumab
- Benralizumab Arm 3 (Experimental): Benralizumab Dose B regimen A until Week 12, Dose B regimen A until Week 24, and Dose B regimen B during the extension period until Week 52 (n=30)
  Interventions: Biological: Benralizumab
- Benralizumab Arm 4 (Experimental): Benralizumab Dose B regimen A until Week 12, Dose B regimen A until Week 24, and Dose B regimen A during the extension period until Week 52 (n=30)
  Interventions: Biological: Benralizumab
- Placebo and Benralizumab (Experimental): Placebo regimen A until Week 24, benralizumab Dose B regiment A until Week 36, and Dose B regimen B until Week 52 (n=40).
  Interventions: Biological: Placebo and Benralizumab

INTERVENTIONS:
Biological: Benralizumab — 2 induction doses of benralizumab (dose A and B) compared to placebo, and a comparison of maintenance dosing regimens (B vs A) in the 28-week extension period.
  Other Names: Benralizumab, Benra, Fasenra
  Arms: Benralizumab Arm 1; Benralizumab Arm 2; Benralizumab Arm 3; Benralizumab Arm 4
Biological: Placebo and Benralizumab — 2 induction doses of benralizumab (dose A and B) compared to placebo, and a comparison of maintenance dosing regimens (B vs A) in the 28-week extension period.
  Other Names: Benralizumab, Benra, Fasenra
  Arms: Placebo and Benralizumab

SUMMARY:
The purpose of this study is to investigate the use of benralizumab is effective in the treatment of chronic spontaneous urticaria (CSU) who are symptomatic despite the use of antihistamines.

DETAILED DESCRIPTION:
The aim of this study is to investigate the use of benralizumab as treatment for patients with chronic spontaneous urticaria (CSU) who are symptomatic despite the use of antihistamines. It is proposed that benralizumab will deplete eosinophils and basophils from affected skin, improve symptoms of CSU, and improve CSU-related quality of life. This Phase 2b study is designed to evaluate induction and maintenance dosing regimens.

ELIGIBILITY:
Inclusion Criteria:

Informed Consent/Age/Gender

1. Provision of the signed and dated written informed consent of the participant prior to any mandatory study-specific procedures, sampling, and analyses.
2. Adult participants≥18 years of age at the time of signing the Informed Consent Form (ICF).

   Type of Participants and Disease
3. Physician-confirmed diagnosis of CSU (also known as chronic idiopathic urticaria) for at least 6 months prior to screening (Visit 1).
4. Presence of pruritus and wheals for at least 6 consecutive weeks prior to screening (Visit 1), despite receiving standard of care, which may include second generation H1 antihistamines (at approved or up to 4-times approved doses) as monotherapy or in combination with LTRAs and/or H2 blockers.
5. Symptomatic during run-in, defined by the following:

   1. UAS7 total score of ≥ 16 with an ISS7 of ≥ 8, during the 7 days prior to randomisation (Visit 2)
   2. In-clinic UAS total score of ≥ 4 on at least one of the screening days.
6. Willing to use a second-generation H1 antihistamine at the approved dose and as monotherapy from the screening visit (Visit 1) until the end of the study.
7. Participants must complete daily PRO assessments and meet the following compliance criteria:

   1. Complete at least 80% of daily PRO assessments between Visit 1 and Visit 2 and
   2. Complete at least 6 of 7 daily PRO assessments in the 7 days prior to Visit 2.
8. Compliance with the locally-approved dose of antihistamine, maintained at randomisation.

   Reproduction
9. Females of childbearing potential (FOCBP) must agree to use a highly effective method of birth control (confirmed by the Investigator) from randomisation, throughout the study duration, and within12 weeks after last dose of IP and have a negative serum pregnancy test result on Visit 1. Highly effective methods of birth control include:

   1. Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal.
   2. Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, or implantable.
   3. Intrauterine device.
   4. Intrauterine hormone-releasing system.
   5. Bilateral tubal occlusion or ligation.
   6. Sexual abstinence, ie, refraining from heterosexual intercourse (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant).
   7. Vasectomised sexual partner (provided that partner is the sole sexual partner of the FOCBP study participant and that the vasectomised partner has received medical assessment of the surgical success).
10. Females not of childbearing potential are defined as Females who are either permanently sterilised (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or who are postmenopausal. Females will be considered postmenopausal if they have been amenorrhoeic for≥12 months prior to the planned date of randomisation without an alternative medical cause. The following age-specific requirements apply:

    1. Females<50 years old will be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and follicle-stimulating hormone (FSH) levels in the postmenopausal range. Until FSH is documented to be within menopausal range, the participant should be treated as a FOCBP.
    2. Females≥50 years old will be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.

Exclusion Criteria:

Medical Conditions

1. Participants with predominant inducible urticaria, ie, urticaria that is predominantly due to a clearly defined stimulus (eg, pressure [dermographism], delayed pressure, cold, heat, sunlight, vibration, water, physical exercise, or increased body temperature [cholinergic]).
2. Participants with diseases, other than chronic urticaria, with urticaria or angioedema symptoms such as urticaria vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa) and hereditary or acquired angioedema (eg, due to C1-inhibitor deficiency). Additionally, any other skin disease associated with chronic itching and/or skin lesions that, in the investigators opinion, might influence the study evaluations and results (eg, atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, etc.).
3. Current malignancy, or history of malignancy, with the exception of: (a) Participants who have had basal cell carcinoma, localised squamous cell carcinoma of the skin, or in situ carcinoma of the cervix are eligible provided that the participant is in remission and curative therapy was completed at least 12 months prior to the date informed consent, was obtained. (b) Participants who have had other malignancies are eligible provided that the participant is in remission and curative therapy was completed at least 5 years prior to the date informed consent, was obtained.
4. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could: (a) Affect the safety of the participant throughout the study (b) Influence the findings of the studies or their interpretations (c) Impede the participant's ability to complete the entire duration of study.
5. History of anaphylaxis to any biologic therapy or vaccine.
6. A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with,or has failed to respond to standard of care therapy.
7. Any clinically significant abnormal findings in physical examination, vital signs, haematology, clinical chemistry, or urinalysis during screening/run-in period which, in the opinion of the Investigator, may put the participant at risk because of his/her participation in the study, or may influence the results of the study, or the participant's ability to complete entire duration of the study.
8. Current active liver disease:

   1. Chronic stable hepatitis B andC (including positive testing for hepatitis B surface antigen [HBsAg] or hepatitis C antibody), or other stable chronic liver disease are acceptable if participant otherwise meets eligibility criteria. Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice, or cirrhosis.
   2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level≥3 times the upper limit of normal (ULN), confirmed by repeated testing during the run-in period. Transient increase of AST/ALT level that resolves by the time of randomisationis acceptable if in the Investigator's opinion the participant does not have an active liver disease and meets other eligibility criteria.
9. A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test. Prior/concomitant Therapy
10. Use of immunosuppressive medication, including, but not limited to: methotrexate, cyclosporine, azathioprine, topical and systemic corticosteroids within 4 weeks or 5 half-lives prior to the date informed consent is obtained, whichever is longer.
11. Known history of allergy or reaction to any component of the IP formulation Other
12. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained
13. Receipt of any marketed (eg, omalizumab) or investigational biologic within 4 months or 5 half-lives prior to the date informed consent is obtained, whichever is longer.
14. Receipt of live attenuated vaccines 30 days prior to the date of randomisation
15. Receipt of any investigational nonbiologic within 30 days or 5 half-lives prior to the date informed consent is obtained, whichever is longer
16. Previously received benralizumab (MEDI-563, FASENRA)
17. Change to allergen immunotherapy or new allergen immunotherapy within 30 days prior to the date of informed consent and anticipated changes in immunotherapy throughout the study
18. Planned elective major surgical procedures during the conduct of the study
19. Previous randomization in the present study
20. Concurrent enrollment in another clinical trial
21. AstraZeneca staff involved in the planning and/or conduct of the study
22. For Females only: Currently pregnant, breastfeeding, or lactating Females (a) A serum pregnancy test will be done for FOCBP at Visit 1 and a urine pregnancy test must be performed for FOCBP at each treatment visit prior to IP administration. A positive urine test result must be confirmed with a serum pregnancy test. If serum test is positive, the participant should be excluded.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Altrichter, MD, Principal Investigator — Charite Universitaetsmedizin Berlin - Campus Charite Mitte
Locations (34):
- United States (11):
  - Research Site, Scottsdale, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Newport Beach, California
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Ypsilanti, Michigan
  - Research Site, Cincinnati, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Austin, Texas
- Bulgaria (4):
  - Research Site, Haskovo
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
- Germany (3):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Leipzig
- Japan (5):
  - Research Site, Hiroshima
  - Research Site, Kamimashikigun,
  - Research Site, Kawasaki-shi
  - Research Site, Kobe
  - Research Site, Sakaishi
- Poland (5):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, Seoul, South Korea
- Spain (5):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Manises

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: ARROYO Patient Brochure — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3259C00001&attachmentIdentifier=0924ff6b-5f3f-4ede-b463-6002e8ad52cb&fileName=AZ_ARROYO_Patient_Brochure_V02Global(en).pdf&versionIdentifier=
- See also: ARROYO Patient Flyer — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3259C00001&attachmentIdentifier=e69cb285-dbb3-4153-b064-f8de4ea8cb85&fileName=AZ_ARROYO_Patient_Flyer_V02Global(en).pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3259C00001&attachmentIdentifier=01965dc3-e23c-4c2f-8254-d3fb97e1059b&fileName=D3259C00001_Synoptic_Clinical_Study_Report_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2b, randomized, double-blind study was conducted in participants with chronic spontaneous urticaria (CSU) who were symptomatic despite the use of antihistamines at 46 study centers in Bulgaria, Germany, Japan, Korea, Poland, Spain, and United States of America between 27 October 2020 and 28 March 2023. The study was terminated early by the sponsor as primary results did not support the continued development of benralizumab for the indication of CSU.
Pre-assignment Details: The study had a run-in period (10 days to 4 weeks), followed by a double-blind treatment period (24 weeks) and extension period (28 weeks). A total of 155 participants were randomized and treated in this study.
Groups:
- Double-blind Then Extension Period: Benralizumab 30 mg Q4W: Participants were randomized to receive benralizumab 30 milligram (mg) subcutaneous (SC) injection every 4 weeks (Q4W) until Week 24 in the double-blind treatment period and then 30 mg Q4W during the extension period until Week 52.
- Double-blind Then Extension Period: Benralizumab 30 mg Q8W: Participants were randomized to receive benralizumab 30 mg SC injection Q4W until Week 24 in the double-blind treatment period and then 30 mg every 8 weeks (Q8W) during the extension period until Week 52.
- Double-blind Then Extension Period: Benralizumab 60 mg Q4W: Participants were randomized to receive benralizumab 60 mg SC injection Q4W until Week 12 and then 30 mg Q4W until Week 24 in the double-blind treatment period followed by 30 mg Q4W during the extension period until Week 52.
- Double-blind Then Extension Period: Benralizumab 60 mg Q8W: Participants were randomized to receive benralizumab 60 mg SC injection Q4W until Week 12 and then 30 mg Q4W until Week 24 in the double-blind treatment period followed by 30 mg Q8W during the extension period until Week 52.
- Double-blind Then Extension Period: Placebo: Participants were randomized to receive placebo matching with benralizumab Q4W until Week 24 in the double-blind treatment period followed by benralizumab 30 mg SC injection Q4W until Week 36 and then 30 mg Q8W until Week 52.
Period: Overall Study
Arm/Group | Double-blind Then Extension Period: Benralizumab 30 mg Q4W | Double-blind Then Extension Period: Benralizumab 30 mg Q8W | Double-blind Then Extension Period: Benralizumab 60 mg Q4W | Double-blind Then Extension Period: Benralizumab 60 mg Q8W | Double-blind Then Extension Period: Placebo
Started | 30 | 29 | 28 | 28 | 40
Completed the Treatment Period | 26 | 27 | 25 | 28 | 37
Entered Extension Period | 24 | 26 | 25 | 28 | 37
Completed | 16 | 21 | 20 | 23 | 24
Not Completed | 14 | 8 | 8 | 5 | 16
Not completed — Adverse Event | 1 | 3 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 3 | 1 | 2 | 4 | 5
Not completed — Withdrawal by Subject | 8 | 3 | 5 | 1 | 9
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug, irrespective of their protocol adherence and continued participation in the study.
Groups:
- Benralizumab 30 mg: Participants were randomized to receive benralizumab 30 mg SC injection Q4W until Week 24 in the double-blind treatment period and then 30 mg Q4W or Q8W during the extension period until Week 52.
- Benralizumab 60 mg: Participants were randomized to receive benralizumab 60 mg SC injection Q4W until Week 12 and then 30 mg Q4W until Week 24 in the double-blind treatment period followed by 30 mg Q4W or Q8W during the extension period until Week 52.
- Placebo: Participants were randomized to receive placebo matching with benralizumab Q4W until Week 24 in the double-blind treatment period followed by benralizumab 30 mg SC injection Q4W until Week 36 and then 30 mg Q8W until Week 52.
- Total: Total of all reporting groups
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo | Total
Number analyzed (Participants) | 59 | 56 | 40 | 155
Age, Customized [Count of Participants; unit: Participants]
  <35 years | 11 | 15 | 8 | 34
  >=35 to <=55 years | 32 | 25 | 22 | 79
  >55 years | 16 | 16 | 10 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 45 | 25 | 114
  Male | 15 | 11 | 15 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 46 | 42 | 30 | 118
  Asian | 12 | 12 | 8 | 32
  Black or African American | 1 | 2 | 0 | 3
  Not reported | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 4 | 10
  Not Hispanic or Latino | 57 | 52 | 36 | 145

OUTCOME MEASURES:

1. Primary Outcome: Least Square (LS) Mean Change From Baseline in Itch Severity Score Over 7 Days (ISS7) at Week 12
Description: The urticaria participant daily diary (UPDD) was completed twice daily (morning and evening) to capture key measures of urticaria disease activity including the itch severity score (ISS). The ISS represents severity on a scale ranging from 0 to 3 (where 0= none, 1= mild, 2= moderate and 3= severe). The ISS7 is the sum of ISS for the previous 7 days. The ISS7 represents itch severity on a scale ranging from 0 (minimum) to 21 (maximum). Higher scores indicate greater intensity of itch. Baseline was defined as the sum of the daily scores for the 7 days prior to the day of randomization.
Time Frame: Baseline (Day -1) and Week 12
Population: The FAS included all randomized participants who received at least 1 dose of study drug, irrespective of their protocol adherence and continued participation in the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 37
units on a scale | -7.50 [-8.94 to -6.05] | -8.28 [-9.76 to -6.80] | -6.49 [-8.24 to -4.74]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.3824, Mixed-effect model for repeated measures — Change from baseline in ISS7 at Week 12= Treatment + baseline ISS7 + region (Europe, North America, Asia) + visit + treatment by visit; LS mean difference = -1.01, 95% CI 2-sided [-3.28 to 1.26]
Statistical Analysis 2: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.1244, Mixed-effect model for repeated measures — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -1.79, 95% CI 2-sided [-4.09 to 0.50]

2. Secondary Outcome: LS Mean Change From Baseline in Urticaria Activity Score Over 7 Days (UAS7) at Weeks 12 and 24
Description: The UPDD was completed twice daily (morning and evening) to capture key measures of urticaria disease activity including the UAS7. Participants were asked to document the number of hives they experienced on a scale ranging from 0 to 3 (where 0= none, 1= mild [1 - 6 hives/12 hour], 2= moderate [7 - 12 hives/12 hour] and 3= intense [(> 12 hives/12 hour]). The UAS7 is the sum of UAS for the previous 7 days, that is, the sum of ISS7 and HSS7. The UAS7 represents urticaria severity on a scale from 0 (minimum) to 42 (maximum). Higher scores indicate greater severity of urticaria symptoms. Baseline was defined as the sum of the daily scores for the 7 days prior to the day of randomization.
Time Frame: Baseline (Day -1) and Weeks 12 and 24
Population: The FAS included all randomized participants who received at least 1 dose of study drug, irrespective of their protocol adherence and continued participation in the study. Participants with data at baseline and each time point were analyzed. The overall number analyzed included those with data at baseline and at least 1 of the reported time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 55 | 53 | 37
units on a scale
  Week 12: number analyzed (Participants) | 55 | 52 | 37
  Week 12 | -14.48 [-17.58 to -11.38] | -16.77 [-19.94 to -13.59] | -12.41 [-16.17 to -8.65]
  Week 24: number analyzed (Participants) | 52 | 53 | 36
  Week 24 | -17.99 [-21.29 to -14.68] | -19.17 [-22.51 to -15.83] | -15.43 [-19.43 to -11.44]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.4016, Mixed-effect model for repeated measures — Change from baseline in UAS7 at Week 12= Treatment + baseline UAS7 + region (Europe, North America, Asia) + visit + treatment by visit; LS mean difference = -2.07, 95% CI 2-sided [-6.95 to 2.80]
Statistical Analysis 2: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.0819, Mixed-effect model for repeated measures — [p-value comment as in outcome 2, analysis 1]; LS mean difference = -4.36, 95% CI 2-sided [-9.28 to 0.56]
Statistical Analysis 3: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.3314, Mixed-effect model for repeated measures — Change from baseline in UAS7 at Week 24= Treatment + baseline UAS7 + region (Europe, North America, Asia) + visit + treatment by visit; LS mean difference = -2.56, 95% CI 2-sided [-7.74 to 2.63]
Statistical Analysis 4: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.1582, Mixed-effect model for repeated measures — [p-value comment as in outcome 2, analysis 3]; LS mean difference = -3.74, 95% CI 2-sided [-8.95 to 1.47]

3. Secondary Outcome: LS Mean Change From Baseline in ISS7 at Week 24
Description: The UPDD was completed twice daily (morning and evening) to capture key measures of urticaria disease activity including the ISS. The ISS represents severity on a scale ranging from 0 to 3 (where 0= none, 1= mild, 2= moderate and 3= severe). The ISS7 is the sum of ISS for the previous 7 days. The ISS7 represents itch severity on a scale ranging from 0 (minimum) to 21 (maximum). Higher scores indicate greater intensity of itch. Baseline was defined as the sum of the daily scores for the 7 days prior to the day of randomization.
Time Frame: Baseline (Day -1) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 52 | 53 | 36
units on a scale | -9.19 [-10.77 to -7.61] | -9.33 [-10.93 to -7.73] | -7.57 [-9.48 to -5.66]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.1995, Mixed-effect model for repeated measures — Change from baseline in ISS7 at Week 24= Treatment + baseline ISS7 + region (Europe, North America, Asia) + visit + treatment by visit; LS mean difference = -1.62, 95% CI 2-sided [-4.10 to 0.86]
Statistical Analysis 2: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.1654, Mixed-effect model for repeated measures — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -1.76, 95% CI 2-sided [-4.25 to 0.73]

4. Secondary Outcome: Percentage of Responders at Weeks 12 and 24
Description: Responder was defined as a participant whose condition was considered clinically well controlled with UAS7 <=6 at specific time points. The UAS7 is the sum of UAS for the previous 7 days, that is, the sum of ISS7 and HSS7. The UAS7 represents urticaria severity on a scale from 0 (minimum) to 42 (maximum). Higher scores indicate greater severity of urticaria symptoms.
Time Frame: Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 59 | 56 | 40
percentage of participants
  Week 12 | 22.0 | 21.4 | 10.0
  Week 24 | 28.8 | 37.5 | 27.5
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.1373, Regression, Logistic — Week 12: Estimates included treatment group, region (Europe, North America, Asia) and baseline UAS7; percentage difference = 11.72, 95% CI 2-sided [-2.37 to 25.82]
Statistical Analysis 2: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.1697, Regression, Logistic — Week 12: Estimates included treatment group, region (Europe, North America, Asia) and baseline UAS7; percentage difference = 10.73, 95% CI 2-sided [-3.42 to 24.88]
Statistical Analysis 3: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.9105, Regression, Logistic — Week 24: Estimates included treatment group, region (Europe, North America, Asia) and baseline UAS7; percentage difference = 1.03, 95% CI 2-sided [-16.90 to 18.96]
Statistical Analysis 4: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.3389, Regression, Logistic — Week 24: Estimates included treatment group, region (Europe, North America, Asia) and baseline UAS7; percentage difference = 9.27, 95% CI 2-sided [-9.37 to 27.90]

5. Secondary Outcome: LS Mean Change From Baseline in Hives Severity Score Over 7 Days (HSS7) at Weeks 12 and 24
Description: The UPDD was completed twice daily (morning and evening) to capture key measures of urticaria disease activity including the HSS7. Participants were asked to document the number of hives they experienced on a scale ranging from 0 to 3 (where 0= none, 1= mild [1 - 6 hives/12 hour], 2= moderate [7 - 12 hives/12 hour] and 3= intense [(> 12 hives/12 hour]). The HSS7 is the sum of hives severity score for the previous 7 days. The HSS7 represents hives severity on a scale from 0 (minimum) to 21 (maximum). Higher scores indicate greater intensity of hives. Baseline was defined as the sum of the daily scores for the 7 days prior to the day of randomization.
Time Frame: Baseline (Day -1) and Weeks 12 and 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 55 | 53 | 37
units on a scale
  Week 12: number analyzed (Participants) | 55 | 52 | 37
  Week 12 | -7.03 [-8.84 to -5.22] | -8.47 [-10.32 to -6.62] | -5.87 [-8.06 to -3.68]
  Week 24: number analyzed (Participants) | 52 | 53 | 36
  Week 24 | -8.88 [-10.76 to -7.00] | -9.81 [-11.71 to -7.91] | -7.82 [-10.09 to -5.54]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.4203, Mixed-effect model for repeated measures — Change from baseline in HSS7 at Week 12= Treatment + baseline HSS7 + region (Europe, North America, Asia) + visit + treatment by visit; LS mean difference = -1.16, 95% CI 2-sided [-4.00 to 1.68]
Statistical Analysis 2: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.0754, Mixed-effect model for repeated measures — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -2.60, 95% CI 2-sided [-5.46 to 0.27]
Statistical Analysis 3: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.4772, Mixed-effect model for repeated measures — Change from baseline in HSS7 at Week 24= Treatment + baseline HSS7 + region (Europe, North America, Asia) + visit + treatment by visit; LS mean difference = -1.06, 95% CI 2-sided [-4.01 to 1.89]
Statistical Analysis 4: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.1851, Mixed-effect model for repeated measures — [p-value comment as in outcome 5, analysis 3]; LS mean difference = -2.00, 95% CI 2-sided [-4.96 to 0.97]

6. Secondary Outcome: Time to >=5-Point Decrease in ISS7
Description: The time to >=5-point decrease (clinically relevant decrease) in ISS7 was reported. The ISS7 is the sum of ISS for the previous 7 days. The ISS7 represents itch severity on a scale ranging from 0 (minimum) to 21 (maximum). Higher scores indicate greater intensity of itch.
Time Frame: From Baseline (Day -1) up to Week 24
Population: The FAS included all randomized participants who received at least 1 dose of study drug, irrespective of their protocol adherence and continued participation in the study. Only participants with at least 1 >=5-point decrease in ISS7 are analyzed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 48 | 50 | 33
weeks | 3.0 [2.0 to 5.0] | 2.0 [2.0 to 3.0] | 8.0 [3.0 to 11.0]

7. Secondary Outcome: Percentage of Participants With Complete UAS7 Response at Weeks 12 and 24
Description: Complete response was defined as participants with UAS7= 0 at specific time points. The UAS7 is the sum of UAS for the previous 7 days, that is, the sum of ISS7 and HSS7. The UAS7 represents urticaria severity on a scale from 0 (minimum) to 42 (maximum). Higher scores indicate greater severity of urticaria symptoms.
Time Frame: Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 59 | 56 | 40
percentage of participants
  Week 12 | 11.9 | 7.1 | 10.0
  Week 24 | 16.9 | 21.4 | 20.0
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.9678, Regression, Logistic — Week 12: Estimates included treatment group, region (Europe, North America, Asia) and baseline UAS7
Statistical Analysis 2: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.3689, Regression, Logistic — Week 12: Estimates included treatment group, region (Europe, North America, Asia) and baseline UAS7
Statistical Analysis 3: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.6624, Regression, Logistic — Week 24: Estimates included treatment group, region (Europe, North America, Asia) and baseline UAS7; percentage difference = -3.43, 95% CI 2-sided [-18.96 to 12.11]
Statistical Analysis 4: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.9726, Regression, Logistic — Week 24: Estimates included treatment group, region (Europe, North America, Asia) and baseline UAS7; percentage difference = 0.28, 95% CI 2-sided [-15.84 to 16.40]

8. Secondary Outcome: Mean Percentage of Angioedema-Free Days Over the Past 7 Days at Weeks 12 and 24
Description: The UPDD included a daily yes/no question asking whether the participant experienced angioedema during the past 24 hours. If yes, the participant was asked a follow-up question about how they treated the swelling. The percentage of angioedema-free days was calculated over the past 7 days by (number of angioedema-free days/number of non-missing responses) x 100.
Time Frame: Weeks 12 and 24
Population: The FAS included all randomized participants who received at least 1 dose of study drug, irrespective of their protocol adherence and continued participation in the study. Only participants with angioedema at baseline or history of angioedema are analyzed.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 36 | 28 | 22
percentage of days
  Week 12: number analyzed (Participants) | 36 | 27 | 22
  Week 12 | 77.50 (35.990) | 85.63 (32.435) | 81.93 (34.548)
  Week 24: number analyzed (Participants) | 32 | 28 | 20
  Week 24 | 78.50 (36.992) | 91.33 (27.032) | 86.79 (31.798)

9. Secondary Outcome: LS Mean Change From Baseline in Urticaria Control Test (UCT) at Weeks 12 and 24
Description: Urticaria disease control was assessed by the UCT using the electronic participant-reported outcome device. The UCT has a retrospective approach using a recall period of 4 weeks and responses on 5-point Likert scales with score ranging from 0 to 4 for each question. Subsequently, the scores for all 4 questions were summed up. The UCT scale range from 0 (minimum) to 16 (maximum). Higher scores indicate better disease control.
Time Frame: Baseline (Day -1) and Weeks 12 and 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 38
units on a scale
  Week 12: number analyzed (Participants) | 55 | 51 | 38
  Week 12 | 4.74 [3.71 to 5.76] | 6.11 [5.05 to 7.17] | 5.02 [3.78 to 6.26]
  Week 24: number analyzed (Participants) | 51 | 52 | 37
  Week 24 | 5.24 [4.04 to 6.45] | 6.87 [5.65 to 8.09] | 5.88 [4.44 to 7.32]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.7256, Mixed-effect model for repeated measures — Change from baseline in UCT at Week 12= Treatment + baseline UCT + region (Europe, North America, Asia) + visit + treatment by visit; LS mean difference = -0.29, 95% CI 2-sided [-1.90 to 1.32]
Statistical Analysis 2: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.1890, Mixed-effect model for repeated measures — [p-value comment as in outcome 9, analysis 1]; LS mean difference = 1.09, 95% CI 2-sided [-0.54 to 2.72]
Statistical Analysis 3: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.5048, Mixed-effect model for repeated measures — Change from baseline in UCT at Week 24= Treatment + baseline UCT + region (Europe, North America, Asia) + visit + treatment by visit; LS mean difference = -0.63, 95% CI 2-sided [-2.51 to 1.24]
Statistical Analysis 4: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.2991, Mixed-effect model for repeated measures — [p-value comment as in outcome 9, analysis 3]; LS mean difference = 0.99, 95% CI 2-sided [-0.89 to 2.88]

10. Secondary Outcome: LS Mean Change From Baseline in Chronic Urticaria Quality of Life Questionnaire (CU-Q2oL) at Weeks 12 and 24
Description: The CU-Q2oL is a 23-item assessment of CSU-specific health-related quality of life. Participants were asked to rate their CSU symptoms and the impact of their symptoms over the last 2 weeks on several domains: pruritus, swelling, impact on life activities, sleep problems, limits, and looks. The questions were scored as 1= not at all, 2= a little, 3= moderately, 4= very much, 5= extremely. The scores were transformed into percentages of the maximum possible score. The CU-Q2oL scale range from 0 (minimum) to 100 (maximum). Higher scores indicate greater impact of urticaria on health-related quality of life.
Time Frame: Baseline (Day -1) and Weeks 12 and 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 38
units on a scale
  Week 12: number analyzed (Participants) | 55 | 51 | 38
  Week 12 | -16.47 [-20.10 to -12.84] | -20.34 [-24.09 to -16.60] | -18.10 [-22.46 to -13.74]
  Week 24: number analyzed (Participants) | 51 | 52 | 37
  Week 24 | -17.60 [-21.81 to -13.40] | -22.11 [-26.38 to -17.84] | -19.07 [-24.09 to -14.05]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.5704, Mixed-effect model for repeated measures — Change from baseline in CU-Q2oL at Week 12= Treatment + baseline CU-Q2oL + region (Europe, North America, Asia) + visit + treatment by visit; LS mean difference = 1.63, 95% CI 2-sided [-4.05 to 7.32]
Statistical Analysis 2: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.4416, Mixed-effect model for repeated measures — [p-value comment as in outcome 10, analysis 1]; LS mean difference = -2.24, 95% CI 2-sided [-7.98 to 3.50]
Statistical Analysis 3: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.6591, Mixed-effect model for repeated measures — Change from baseline in CU-Q2oL at Week 24= Treatment + baseline CU-Q2oL + region (Europe, North America, Asia) + visit + treatment by visit; LS mean difference = 1.47, 95% CI 2-sided [-5.09 to 8.02]
Statistical Analysis 4: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.3624, Mixed-effect model for repeated measures — [p-value comment as in outcome 10, analysis 3]; LS mean difference = -3.04, 95% CI 2-sided [-9.62 to 3.54]

11. Secondary Outcome: LS Mean Change From Baseline in Dermatology Life Quality Index (DLQI) at Weeks 12 and 24
Description: The DLQI is a 10-item assessment of dermatology-specific health-related quality of life. Participants were asked to rate their symptoms and the impact of their symptoms over the last week on several domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The questions (except question 7) were scored on a 4-point Likert scale: 0= not at all, 1= a little, 2= a lot, 3= very much. Scoring question 7, the first part asked: 'Over the last week, has your skin prevented you from working or studying?' Scoring was for response of 0= not relevant and 3= yes. If response was 'no', a further question was asked: 'How much has your skin been a problem at work or studying', and scored as: 0= not at all, 1= a little, 2= a lot. The DLQI was calculated by summing the score of each question. The DLQI scale range from 0 (minimum) to 30 (maximum). Higher scores indicate greater impact on participant's life.
Time Frame: Baseline (Day -1) and Weeks 12 and 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 38
units on a scale
  Week 12: number analyzed (Participants) | 55 | 51 | 38
  Week 12 | -7.58 [-9.18 to -5.98] | -9.31 [-10.96 to -7.66] | -8.06 [-9.98 to -6.14]
  Week 24: number analyzed (Participants) | 51 | 52 | 37
  Week 24 | -8.13 [-9.84 to -6.42] | -10.25 [-11.98 to -8.51] | -9.37 [-11.41 to -7.33]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.7037, Mixed-effect model for repeated measures — Change from baseline in DLQI at Week 12= Treatment + baseline DLQI + region (Europe, North America, Asia) + visit + treatment by visit; LS mean difference = 0.48, 95% CI 2-sided [-2.02 to 2.98]
Statistical Analysis 2: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.3320, Mixed-effect model for repeated measures — [p-value comment as in outcome 11, analysis 1]; LS mean difference = -1.25, 95% CI 2-sided [-3.78 to 1.29]
Statistical Analysis 3: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.3590, Mixed-effect model for repeated measures — Change from baseline in DLQI at Week 24= Treatment + baseline DLQI + region (Europe, North America, Asia) + visit + treatment by visit; LS mean difference = 1.24, 95% CI 2-sided [-1.42 to 3.90]
Statistical Analysis 4: Comparison: Benralizumab 60 mg vs Placebo; Test type: Superiority; p = 0.5175, Mixed-effect model for repeated measures — [p-value comment as in outcome 11, analysis 3]; LS mean difference = -0.88, 95% CI 2-sided [-3.56 to 1.80]

12. Secondary Outcome: Serum Concentration of Benralizumab
Description: Blood samples were collected to determine the serum concentration of benralizumab.
Time Frame: Pre-dose on Weeks 4, 12 and 24
Population: The Pharmacokinetic (PK) analysis set included all participants who received study drug and from whom PK blood samples were assumed not to be affected by factors such as protocol violations and who had at least 1 quantifiable serum PK observation post first dose. Placebo group samples were not analyzed at Weeks 4 and 12 as they have not received benralizumab in double-blind treatment period.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 55 | 54 | 34
nanogram per milliliter (ng/mL)
  Week 4: number analyzed (Participants) | 55 | 54 | 0
  Week 4 | 990.515 (448.6799) | 2167.606 (991.7509) |
  Week 12: number analyzed (Participants) | 53 | 52 | 0
  Week 12 | 1321.373 (740.5070) | 3145.352 (1577.6726) |
  Week 24: number analyzed (Participants) | 47 | 49 | 34
  Week 24 | 1372.806 (883.5830) | 1638.810 (946.9466) | NA (NA) — Below the lower limit of quantification (LLOQ). The LLOQ is 3.86 ng/mL.

13. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response to Benralizumab
Description: Blood samples were measured for the presence of ADAs for benralizumab using validated assays. The ADA incidence (treatment-emergent ADA positive) was defined as ADA negative at baseline and post-baseline ADA positive, or ADA positive at baseline and boosted the pre-existing titre by > 4-fold during the study period. Persistently positive was defined as ADA negative at baseline and positive at >= 2 post-baseline assessments (with >= 16 weeks between first and last positive) or positive at last post-baseline assessment. Transiently positive was defined as ADA negative at baseline, having at least 1 post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive. The median of maximum titres was calculated based on the maximum titre for each ADA positive participant within each treatment group (including both baseline and post-baseline measurements).
Time Frame: Pre-dose on Weeks 12 and 24
Population: The Safety analysis set included all participants who received at least 1 dose of study drug. Participants with data at baseline and at least 1 post baseline sample were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Benralizumab 60 mg | Placebo
Number analyzed (Participants) | 59 | 56 | 40
Participants
  ADA prevalence | 18 | 13 | 4
  ADA negative (both baseline and post-baseline negative): number analyzed (Participants) | 54 | 54 | 37
  ADA negative (both baseline and post-baseline negative) | 37 | 41 | 33
  Only baseline positive: number analyzed (Participants) | 55 | 55 | 39
  Only baseline positive | 1 | 1 | 0
  Baseline and at least 1 post-baseline positive | 3 | 4 | 0
  ADA incidence: number analyzed (Participants) | 54 | 54 | 37
  ADA incidence | 15 | 10 | 4
  ADA persistently positive: number analyzed (Participants) | 54 | 54 | 37
  ADA persistently positive | 10 | 4 | 4
  ADA transiently positive: number analyzed (Participants) | 54 | 54 | 37
  ADA transiently positive | 5 | 5 | 0
  ADA positive with maximum titre > median of maximum titres | 8 | 5 | 1
  ADA positive with maximum titre <= median of maximum titres | 10 | 8 | 3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are reported from the first dose administration up to 30days after the last dose of study drug, a maximum of approximately 57 weeks.
Description: The Safety analysis set included all participants who received at least 1 dose of study drug. Only TEAEs that started or worsened in severity on or after first dose of study drug are reported. TEAEs occurred prior to first dose of study drug are not reported as it was pre-specified to report only TEAEs that started or worsened in severity on or after first dose of study drug.
Groups:
- Double-blind Period: Benralizumab 30 mg Q4W: Participants were randomized to receive benralizumab 30 mg SC injection Q4W until Week 24 in the double-blind treatment period.
- Double-blind Period: Benralizumab 60 mg Q4W: Participants were randomized to receive benralizumab 60 mg SC injection Q4W until Week 12 and then 30 mg Q4W until Week 24 in the double-blind treatment period.
- Double-blind Period: Placebo: Participants were randomized to receive placebo matching with benralizumab Q4W until Week 24 in the double-blind treatment period.
- Extension Period: Benralizumab 30 mg Q4W: Participants were randomized to receive benralizumab 30 mg SC injection Q4W in the extension period until Week 52.
- Extension Period: Benralizumab 30 mg Q8W: Participants were randomized to receive benralizumab 30 mg SC injection Q8W in the extension period until Week 52.
- Extension Period: Placebo to Benralizumab: Participants randomized to placebo in the double-blind period received benralizumab 30 mg SC injection Q4W until Week 36 and then 30 mg Q8W until Week 52 in the extension period.
Arm/Group | Double-blind Period: Benralizumab 30 mg Q4W | Double-blind Period: Benralizumab 60 mg Q4W | Double-blind Period: Placebo | Extension Period: Benralizumab 30 mg Q4W | Extension Period: Benralizumab 30 mg Q8W | Extension Period: Placebo to Benralizumab
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/56 | 0/40 | 0/49 | 0/54 | 0/37
Serious Adverse Events (participants affected / at risk) | 3/59 | 1/56 | 0/40 | 0/49 | 3/54 | 1/37
Other Adverse Events (participants affected / at risk) | 14/59 | 13/56 | 10/40 | 16/49 | 12/54 | 11/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Period: Benralizumab 30 mg Q4W (N=59) | Double-blind Period: Benralizumab 60 mg Q4W (N=56) | Double-blind Period: Placebo (N=40) | Extension Period: Benralizumab 30 mg Q4W (N=49) | Extension Period: Benralizumab 30 mg Q8W (N=54) | Extension Period: Placebo to Benralizumab (N=37)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Period: Benralizumab 30 mg Q4W (N=59) | Double-blind Period: Benralizumab 60 mg Q4W (N=56) | Double-blind Period: Placebo (N=40) | Extension Period: Benralizumab 30 mg Q4W (N=49) | Extension Period: Benralizumab 30 mg Q8W (N=54) | Extension Period: Placebo to Benralizumab (N=37)
COVID-19 (Infections and infestations) | 5 (5) | 5 (5) | 1 (1) | 4 (4) | 4 (4) | 5 (5)
Nasopharyngitis (Infections and infestations) | 1 (2) | 4 (4) | 2 (2) | 5 (7) | 2 (2) | 2 (3)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (6) | 0 (0) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early by the sponsor as the primary analysis results did not support the continued development of benralizumab for the indication of CSU.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/25/NCT04612725/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT04612725/SAP_001.pdf